CLINICAL TRIAL: NCT02384863
Title: The Evaluation and Management of Patients With Acute Chest Pain in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuguo Chen (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government); West China Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Chest Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Henan Provincial People's Hospital (Other); Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yuguo Chen, President-elect, Chinese Society of Emergency Medicine;Director, Chest Pain Center, Qilu Hospital of Shandong University, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: 201502032; ChiCTR-IOQ-14005268 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: Chest Pain; Acute Coronary Syndrome; Cardiac; Emergency Department; Cardiac Testing; Healthcare Utilization; Patient Centered Outcomes; Shared Decision Making; Unnecessary hospital admissions; Decision Aid
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe the characteristics, evaluation, management and outcomes of acute chest pain, and to provide opportunities for future initiatives to improve the emergency care for patients experiencing acute chest pain in China.

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain(pain in the area inferior to the clavicle, superior to the rib arch, and anterior to the bilateral posterior axillary line）;
* Possible Acute Coronary Syndrome;
* Symptoms occurring within last 24 hours;
* Informed consent from patient or next of kin.

Exclusion Criteria:

* Arrhythmia or heart failure not cause by myocardial ischemia;
* Confirmed lung disease without chest pain;
* No onset of symptoms within last 24 hours;
* No written consensus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients attending the emergency department in 7 Chinese grade Ⅲ hospitals
Sampling Method: Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | During hospital stay,an expected average of 7 days

SECONDARY OUTCOMES:
Time between symptom onset and hospital admission | Time interval from symptom onset to arrival at the Emergency Department，an expected median of 9 hours
Major adverse cardiac events (MACE) | 1 year
  Composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization
Cost-Effectiveness Analysis | 1 year
  To study the cost-effectiveness ratios of diagnostic and management strategies for patients with acute chest pain

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, M.D., Ph.D., Study Chair — Qilu Hospital of Shandong University
Locations (7):
- China (7):
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial Hospital, Zhengzhou, Henan
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan